CLINICAL TRIAL: NCT06835348
Title: An Observational, Multicenter Study Evaluating the Safety of ReAl-lifePertuzumab and Trastuzumab Fixed Dose Combination: the RAPID Study
Acronym: GIM30-RAPID
Status: Completed | Type: Observational
Sponsor: Fondazione Oncotech (Other)
Responsible Party: Sponsor
Other Study IDs: GIM30-RAPID
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients with HER-2 positive breast cancer: patients with HER-2 positive breast cancer who have completed concurrent chemotherapy with pertuzumab and trastuzumab administered IV and are currently receiving or will be receiving maintenance therapy with PH FDC SC and have at least 6 cycles of therapy expected with PH FDC SC to conclude pre-established oncological treatment.

SUMMARY:
This is a single arm prospective, observational multi-centre study in patients with HER-2 positive breast cancer who have completed concurrent chemotherapy with pertuzumab and trastuzumab administered IV and are currently receiving or will be receiving maintenance therapy with PH FDC SC and have at least 6 cycles of therapy expected with PH FDC SC to conclude pre-established oncological treatment.

Treatment of the patients will not be determined or assigned by study procedures but will be based on normal clinical practice. Only data available per clinical practice will be collected within this study. The treatment decision must have been taken prior to and irrespective of patient's inclusion in the study.

DETAILED DESCRIPTION:
Primary objective

• The primary objective of the study is to evaluate the safety of pertuzumab and trastuzumab (PH) fixed-dose combination (FDC) for subcutaneous (SC) administration in patients with HER-2 positive breast cancer who have completed concurrent chemotherapy with pertuzumab and trastuzumab administered intravenously (IV) and are currently receiving or will be receiving maintenance therapy with PH FDC SC.

Secondary objectives

The secondary exploratory objectives of the study are:

* To assess the patient's social cost saving by means of a specific questionnaire;
* To assess the patient's health related quality of life (HRQOL).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent of the patient;
* Female and male patients aged ≥ 18 years (no upper limit);
* Patients with HER-2 positive breast cancer, who have completed concurrent chemotherapy with pertuzumab and trastuzumab IV and are currently receiving or will be receiving maintenance therapy with PH FDC SC according to locally approved indication;
* Patients with expected at least 6 cycles of therapy with PH FDC SC to conclude pre-established oncological treatment;

Exclusion Criteria:

* Life expectancy < 6 months;
* Presence of any contraindication with regard to treatment with PH FDC SC as specified in the corresponding Summary of Product Characteristics (SmPCs) approved in Italy;
* Concomitant participation in another interventional or non-interventional trial.
* Patients with less than 6 remaining cycles of therapy with PH FDC SC to conclude pre-established oncological treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with HER-2 positive breast cancer who have completed concurrent chemotherapy with pertuzumab and trastuzumab administered IV and are currently receiving or will be receiving maintenance therapy with PH FDC SC and have at least 6 cycles of therapy expected with PH FDC SC to conclude pre-established oncological treatment.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2024-11-29 (Actual)

PRIMARY OUTCOMES:
Number and percentage of patients with grade 3-4 adverse events (AEs), according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE v5.0). | From enrollment to the end of the study (about 24 months)

SECONDARY OUTCOMES:
Other safety endpoints: number and percentage of patients with any AE, serious AEs, fatal AEs, AEs leading to withdrawal of study drug, adverse events of special interest (AESI, refer to Section 13.1.3 for the list); | From enrollment to the end of the study (about 24 months)
Patient's social cost evaluated by means of estimation of indirect costs (Loss of productivity for patients and caregiver) using a specific questionnaire administered at the Screening, after the third cycle of therapy and at the End of Treatment visit; | From enrollment to the end of the study (about 24 months)
Patient's HRQOL, evaluated by means of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTC QLQ-C30) administered at the Screening, after the third cycle of therapy and at the End of Treatment visit. | From enrollment to the end of the study (about 24 months)

CONTACTS AND LOCATIONS:
Locations (7):
- Italy (7):
  - A.O.R.N. San Giuseppe Moscati, Avellino, AV
  - A.O.R.N. Caserta "Sant'Anna e San Sebastiano", Caserta, CE
  - Istituto Nazionale Tumori "Fondazione G. Pascale", Naples, Naples
  - Irccs - Centro Riferimento Oncologico (C.R.O.) Di Aviano, Aviano, PN
  - IRCCS Istituto Nazionale Tumori Regina Elena, Rome, Rome
  - Fondazione Policlinico Universitario A. Gemelli IRCSS, Rome, Rome
  - ASL Napoli 3 sud - Stabilimento di Pollena " Cav. R. Apicella", Pollena Trocchia

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available